CLINICAL TRIAL: NCT03818854
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Trial of Allogeneic Bone Marrow-derived Human Mesenchymal Stromal Cells (hMSCs) for the Treatment of Acute Respiratory Distress Syndrome
Brief Title: Mesenchymal Stromal Cells For Acute Respiratory Distress Syndrome
Acronym: STAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael A. Matthay (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Harborview Injury Prevention and Research Center (Other); Oregon Health and Science University (Other); Vanderbilt University Medical Center (Other); The University of Texas Health Science Center, Houston (Other); University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Michael A. Matthay, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSF-hMSC-ARDS-P1P2-12
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Human Mesenchymal Stromal Cells; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: For this Phase 2b trial, after informed consent is given, an assignment will be made by computer-generated randomization to administer either hMSCs therapy or placebo with a 1:1 allocation to the hMSCs:placebo arms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Human Mesenchymal Stromal Cells (Experimental): A single dose of 10 million cells/kg predicted body weight (PBW) Allogeneic Bone Marrow-Derived Human Mesenchymal Stromal Cells will administered intravenously over approximately 60-80 minutes.
  Interventions: Biological: Human Mesenchymal Stromal Cells
- Cell Reconstitution Media (Experimental): A single dose of cell reconstitution media (1:1 mix of 5% human serum albumin and 10% Dextran 40) will administered intravenously over approximately 60-80 minutes.
  Interventions: Biological: Cell Reconstitution Media

INTERVENTIONS:
Biological: Human Mesenchymal Stromal Cells — Immediately prior to administration, the study product will be thawed and diluted 1:1 with reconstitution media (1:1 mix of 5% human serum albumin and 10% Dextran 40). Additional reconstitution media is added to a final product volume of 300 mL.
  Other Names: hMSCs
  Arms: Human Mesenchymal Stromal Cells
Biological: Cell Reconstitution Media — 300 mL of reconstitution media (1:1 mix of 5% human serum albumin and 10% Dextran 40)
  Other Names: Placebo
  Arms: Cell Reconstitution Media

SUMMARY:
This is a Phase 2b, randomized, double-blind, placebo-controlled, multi-center study to assess the safety and efficacy of a single dose of Allogeneic Bone Marrow-derived Human Mesenchymal Stromal Cells (hMSCs) infusion in patients with Acute Respiratory Distress Syndrome (ARDS). This study is the extension of the Phase 1 pilot study (NCT01775774) and Phase 2a study (NCT02097641).

DETAILED DESCRIPTION:
This clinical study design is a randomized, double-blinded, placebo-controlled Phase 2b clinical trial using a 10 million cell/kg dose of human Mesenchymal Stromal Cells (hMSCs). Subjects will be randomized in a 1:1 randomization scheme to receive hMSCs or cell reconstitution media (1:1 mix of 5% human serum albumin and 10% Dextran 40) as the placebo; the study will enroll 120 patients who achieve a stable clinical baseline and receive study product (either hMSCs or the placebo).

The Data and Safety Monitoring Board (DSMB) will review adverse outcomes and protocol compliance. A pre-specified interim review will occur after 60 subjects have been enrolled and received study product; enrollment will continue during the DSMB review. All pre-specified clinically important events and unexpected serious adverse events including death during hospitalization up to 60 days will be reported to the DSMB on an ongoing basis; the study will be stopped for a safety evaluation by the DSMB if they have any concerns or if three subjects have pre-specified clinically important events or unexpected serious adverse events except death since death will be common in this critically ill population due the nature of the underlying illness (e.g., ARDS).

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if they meet all of the below criteria within 14 days of initial ICU admission. Criteria 1-3 must all be present within a 24-hour time period and at the time of enrollment:

Acute onset (defined below) of:

1. A need for positive pressure ventilation by an endotracheal or tracheal tube with a PaO2/FiO2 ratio <250 mmHg and ≥5 cm H2O positive end-expiratory airway pressure (PEEP), as per the Berlin Criteria.
2. Bilateral infiltrates consistent with pulmonary edema (defined below) on the frontal chest radiograph, or bilateral ground glass opacities on a chest CT scan.
3. No clinical evidence of left atrial hypertension as a primary explanation for the bilateral pulmonary infiltrates.
4. If the cause of ARDS is trauma, additional inclusion criteria will include ONE of the following relevant risk factors for developing ARDS:

   1. Hypotension (systolic blood pressure[SBP] < 90 mmHg) in the field or in the first 24 h after injury, or
   2. Transfusion of 3 units of blood products in the first 24 hours following injury, or
   3. Meets the new Critical Administration Threshold (CAT) criteria with at least 3 units of blood in one hour, or
   4. Blunt or penetrating torso trauma, or
   5. Long bone fractures, or
   6. The highest level of institutional trauma activation

Exclusion Criteria:

1. Age less than 18 years
2. Greater than 72 hours since first meeting ARDS criteria per the Berlin definition of ARDS
3. Greater than 14 days since initial ICU admission
4. Inability to administer study product within 14 days of ICU admission
5. PaO2/FiO2 ≥ 250 mmHg after consent obtained and before study product is administered
6. Unable to obtain informed consent/no surrogate available
7. Pregnant or lactating
8. In custody of law enforcement officials
9. Burns > 20% of total body surface area
10. WHO Class III or IV pulmonary hypertension
11. History of cancer treatment in the last 2 years except for non-melanotic skin cancers
12. Underlying medical condition for which 6-month mortality is estimated to be > 50%
13. Moribund patient not expected to survive 24 hours
14. Advanced chronic liver disease (Child-Pugh Score > 12)
15. Severe chronic respiratory disease with the use of home oxygen
16. Severe traumatic brain injury - defined as:

    1. A patient who has undergone intracranial neurosurgical intervention for monitoring or therapy (intracranial pressure monitoring, external ventricular drain, craniotomy), or
    2. Intracranial injury by head CT (does not include patients with minimal subarachnoid injury and/or minor skull fracture), or
    3. Post-resuscitation Glasgow Coma Score (GCS) < 9 assessed after sedation interruption, or
    4. Non-survivable head injury as assessed by neurosurgery
17. Evidence of anoxic brain injury
18. History of stroke within the last 3 years
19. No intent/unwillingness to follow lung protective ventilation strategy
20. Currently receiving extracorporeal life support (ECLS) or high-frequency oscillatory ventilation (HFOV)
21. Anticipated extubation within 24 hours of enrollment
22. Clinical evidence of left atrial hypertension as measured by a pulmonary arterial wedge pressure > 18mmHg or left ventricular failure measured by an echocardiogram with a left ventricular ejection fraction less than 40%. Clinical judgement will determine if either of these measurements needs to be carried out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Matthay, MD, Principal Investigator — University of California, San Francisco
Locations (7):
- United States (7):
  - University of California Davis Medical Center, Sacramento, California
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We do not have plan to share IPD data to other researchers.

REFERENCES:
- [Derived] Matthay MA, Zhou H, Sarma A, Alipanah-Lechner N, Hendrickson C, Kornblith LZ, Schreiber M, Zonies D, Khan A, Robinson B, Johnson NJ, Ware LB, Guillamondegui O, Casey J, Moore L, Patel B, Kao L, Wade CE, Fox E, Cox C, Khawanja F, Aguillon Prada R, Hossri S, Callcut R, Albertson T, Delucchi KL, McMillan M, Langelier CR, Pati S, McKenna DH, Leroux C, Calfee CS, Liu KD. Treatment with Allogenic Mesenchymal Stromal Cells for Moderate to Severe Acute Respiratory Distress Syndrome: A Double-Blind, Placebo-controlled, Multi-Center, Phase 2b Clinical Trial (STAT). Am J Respir Crit Care Med. 2025 Jul 29:10.1164/rccm.202411-2254OC. doi: 10.1164/rccm.202411-2254OC. Online ahead of print. PMID 40728562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Started | 59 | 61
Completed | 59 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (14.4) | 57.0 (15.1) | 55.5 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 29 | 49
  Male | 39 | 32 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 26 | 47
  Not Hispanic or Latino | 30 | 31 | 61
  Unknown or Not Reported | 8 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 22 | 32 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  United States | 59 | 61 | 120
COVID positive [Count of Participants; unit: Participants]
  Yes | 56 | 45 | 101
  No | 3 | 16 | 19
Primary Cause of ARDS [Count of Participants; unit: Participants]
  COVID-19 Pneumonia | 56 | 44 | 100
  Non COVID-19 Pneumonia | 0 | 5 | 5
  Sepsis | 1 | 3 | 4
  Trauma | 2 | 5 | 7
  Aspiration | 0 | 3 | 3
  Other | 0 | 1 | 1
Acute Physiology, Age, Chronic Health Evaluation (APACHE) III [Mean (Standard Deviation); unit: units on a scale] — The worst values within 24 hours prior to randomization were calculated for APACHE III score. The range of APACHE III score is from 0 to 299. In APACHE III scoring, the patient's age is worth up to 24, and chronic health history is worth up to 23 points, 17 physiologic variables are measured and may add up to a maximum of an additional 252 points. The higher score, the worse clinical outcome. Population: Data are missing in 5 patients because patients/surrogates refused to release AIDS data.
  units on a scale
    number analyzed (Participants) | 56 | 59 | 115
    (all) | 100.8 (26.0) | 93.6 (26.0) | 97.1 (26.1)
Non-pulmonary Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — The SOFA score comprises of the sum of six organ system components (respiratory, cardiovascular, hepatic, coagulation, renal and neurological) and scores range from 0 to 24 (each component ranges from 0 to 4), with higher values representing a worse organ dysfunction and morbidity.
  units on a scale | 6.9 (3.3) | 6.5 (2.6) | 6.7 (3.0)
Minute Ventilation [Mean (Standard Deviation); unit: liter/min] | 10.0 (2.8) | 9.4 (2.4) | 9.7 (2.6)
PaO2:FiO2 [Mean (Standard Deviation); unit: mmHg] | 152 (44) | 154 (39) | 153 (42)
Lung Injury Score [Mean (Standard Deviation); unit: units on a scale] — Lung Injury Score (LIS) is a validated 4-point score based on chest radiograph findings, PaO2/FiO2 ratio, PEEP and compliance. Scoring is performed for each individual component, and the score is the average of the 4 components. The scores range from 0 to 4, with higher values representing a worse lung injury. Population: Data missing in one patient due to no quadrant value available for lung injury score calculation.
  units on a scale
    number analyzed (Participants) | 58 | 61 | 119
    (all) | 3.2 (0.4) | 3.0 (0.4) | 3.1 (0.4)
Oxygenation Index [Mean (Standard Deviation); unit: cmH20/mmHg] — Oxygenation index calculated as: FiO2 (%) x Mean Airway Pressure (mmHg) / PaO2 (mmHg). The higher value, the worse clinical outcome. Population: Data missing in one patient treated with Cell Reconstitution Media (Placebo) because the patient had pressure support ventilation (PSV), and the oxygenation index was not calculated.
  cmH20/mmHg
    number analyzed (Participants) | 59 | 60 | 119
    (all) | 13.6 (6.6) | 12.1 (4.4) | 12.8 (5.6)
Ventilatory Ratio [Mean (Standard Deviation); unit: ratio] — Ventilatory ratio is a simple bedside measurement of ventilation, which is calculated using the following formula: minute ventilation (ml/min) × PaCO2 (mm Hg)]/(predicted body weight × 100 × 37.5). The higher value, the worse outcome.
  ratio | 2.0 (0.8) | 1.9 (0.6) | 1.9 (0.7)
Angiopoietin 2 (ANG-2) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Some baseline samples were not obtained during the COVID-19 pandemic due to local institutional policies.
  pg/mL
    number analyzed (Participants) | 43 | 45 | 88
    (all) | 3519 [1726 to 7829] | 3755 [2324 to 10158] | 3593 [2191 to 8111]
Interleukin 6 (IL-6) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Some baseline samples were not obtained during the COVID-19 pandemic due to local institutional policies.
  pg/mL
    number analyzed (Participants) | 43 | 45 | 88
    (all) | 56.3 [16.8 to 191.0] | 23.2 [9.7 to 121.2] | 37.1 [11.9 to 183.9]
Interleukin 8 (IL-8) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Some baseline samples were not obtained during the COVID-19 pandemic due to local institutional policies.
  pg/mL
    number analyzed (Participants) | 43 | 45 | 88
    (all) | 14.8 [8.6 to 29.9] | 12.8 [8.3 to 23.8] | 14.2 [8.5 to 26.7]
Receptor for Advanced Glycation Endproducts (RAGE) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Some baseline samples were not obtained during the COVID-19 pandemic due to local institutional policies.
  pg/mL
    number analyzed (Participants) | 43 | 45 | 88
    (all) | 5736 [3245 to 12985] | 6373 [2728 to 12218] | 6229 [2986 to 12547]
Tumor Necrosis Factor Receptor 1 (TNFR-1) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Some baseline samples were not obtained during the COVID-19 pandemic due to local institutional policies.
  pg/mL
    number analyzed (Participants) | 43 | 45 | 88
    (all) | 3492 [2658 to 5819] | 3919 [2576 to 5361] | 3758 [2611 to 5629]
Protein C [Median (Inter-Quartile Range); unit: pg/mL] — Population: Some baseline samples were not obtained during the COVID-19 pandemic due to local institutional policies.
  pg/mL
    number analyzed (Participants) | 42 | 44 | 86
    (all) | 104.3 [75.8 to 133.2] | 99.7 [72.6 to 131.4] | 102.2 [74.5 to 133.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygenation Index (OI)
Description: Change in OI from baseline over the 36 hours (6, 12, 18, 24, 30, 36 hours) following the initiation of the study product infusion. Lower values are considered better.
Time Frame: 36 hours
Population: Missing data are due to various causes: ventilated by PSV mode, not recorded, or expired.
Measure: Median (Inter-Quartile Range); unit: cmH20/mmHg
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
cmH20/mmHg
  6 Hour: number analyzed (Participants) | 57 | 58
  6 Hour | -0.7 [-2.7 to 1.4] | -1.5 [-3.0 to 1.0]
  12 Hour: number analyzed (Participants) | 53 | 55
  12 Hour | 0.8 [-1.6 to 3.5] | -1.1 [-3.9 to 0.9]
  18 Hour: number analyzed (Participants) | 55 | 55
  18 Hour | 0.3 [-3.4 to 3.5] | -1.0 [-4.1 to 2.5]
  24 Hour: number analyzed (Participants) | 52 | 50
  24 Hour | 0.3 [-3.7 to 5.9] | -1.1 [-4.2 to 2.2]
  30 Hour: number analyzed (Participants) | 52 | 50
  30 Hour | 0.8 [-3.3 to 3.8] | -0.7 [-4.0 to 1.0]
  36 Hour: number analyzed (Participants) | 55 | 51
  36 Hour | 0.8 [-3.5 to 5.0] | -1.5 [-3.9 to 0.9]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority — Using the change in oxygenation index over 36 hours from the baseline as the primary outcome with measurements taken at 6 time points, the trial was estimated to have 80% power to detect an effect size difference of 0.43 between the trial arms; p = 0.34, Mixed Models Analysis — The mixed model included the following variables: treatment arm, 6 time-points, sites, pre-defined randomization stratifications and the baseline characteristics with bivariate analyses P < 0.20

2. Secondary Outcome: Acute Lung Injury Score (LIS)
Description: Changes in the 4-point acute lung injury (LIS) score from the baseline to days 1, 2, 3 and 7, or on the last day of positive pressure ventilation prior to day 7. The LIS is a composite 4-point scoring system including the PaO2/FiO2, PEEP, lung compliance, and the extent of infiltrates on the chest X-ray. Each of the four components is categorized from 0 to 4, where a higher number is worse. The total Lung Injury Score is obtained by dividing the aggregate sum by the number of components used.
Time Frame: 7 days
Population: LIS were calculated for patients who were intubated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
score on a scale
  Day 1: number analyzed (Participants) | 52 | 57
  Day 1 | -0.10 (0.41) | -0.10 (0.48)
  Day 2: number analyzed (Participants) | 54 | 55
  Day 2 | -0.07 (0.41) | -0.15 (0.62)
  Day 3: number analyzed (Participants) | 53 | 49
  Day 3 | -0.15 (0.53) | -0.09 (0.57)
  Day 7: number analyzed (Participants) | 38 | 37
  Day 7 | -0.39 (0.69) | -0.21 (0.63)
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change of LIS from the baseline to day 1; Test type: Superiority; p = 0.92, t-test, 2 sided
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change of LIS from the baseline to day 2; Test type: Superiority; p = 0.37, t-test, 2 sided
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change of LIS from the baseline to day 3; Test type: Superiority; p = 0.54, t-test, 2 sided
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change of LIS from the baseline to day 7; Test type: Superiority; p = 0.19, t-test, 2 sided

3. Secondary Outcome: Pulmonary Dead Space Fraction
Description: Pulmonary Dead Space at day 1, 2, 3 and 7. The dead-space fraction is calculated as: (PaCO2 - PeCO2) ÷ PaCO2
Time Frame: 7 days
Population: Due to the COVID-19 pandemic, the master majority of the enrolled patients had COVID-19, and it was not feasible to conduct the pulmonary dead space measurement because if would have increased the risk of spreading the COVID-19 virus to the health care workers, especially the respiratory therapists. Thus, this analysis is not available.
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change of Chest Radiograph Assessment of Pulmonary Edema (RALE Score)
Description: Changes of RALE score at day 1, 2, 3 and 7 from baseline RALE score. To calculate RALE, each radiographic quadrant is scored for extent of consolidation (0-4) and density of opacification (1-3). The product of the consolidation and density scores for each of the four quadrants is summed. The RALE score ranges from 0 (best) to 48 (worst).
Time Frame: 7 days
Population: RALE scores are calculated by the available Chest X-ray photographs.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
score on a scale
  Day 1: number analyzed (Participants) | 33 | 35
  Day 1 | -0.7 [-3.3 to 2.9] | 1.0 [-2.5 to 5.0]
  Day 2: number analyzed (Participants) | 30 | 34
  Day 2 | -1.1 [-5.8 to 4.3] | 1.7 [-2.7 to 4.5]
  Day 3: number analyzed (Participants) | 34 | 33
  Day 3 | -0.5 [-4.7 to 4.3] | 0.0 [-3.4 to 4.0]
  Day 7: number analyzed (Participants) | 31 | 34
  Day 7 | -2.3 [-9.3 to 5.7] | 2.4 [-1.7 to 8.0]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change in RALE scores from the baseline to day 1; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change in RALE scores from the baseline to day 2; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change in RALE scores from the baseline to day 3; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the change in RALE scores from the baseline to day 7; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Ventilator Free-days (VFD) Over 14 Days
Description: Ventilator free-days over 14 days. Defined as the number of days from the time of initiating unassisted breathing to day 14 after study product administration, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 14. If a patient returns to assisted breathing and subsequently achieves unassisted breathing to day 14, VFDs will be counted from the end of the last period of assisted breathing to day 14.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants
  0 day | 44 | 32
  1 - 4 days | 4 | 7
  5 - 9 days | 7 | 12
  10 - 13 days | 4 | 10
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p = 0.01, Regression, Logistic — P-value was given by ordered logistic regression model

6. Secondary Outcome: Ventilator Free-days (VFD) Over 28 Days.
Description: Defined as the number of days from the time of initiating unassisted breathing to day 28 after study product administration, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a patient returns to assisted breathing and subsequently achieves unassisted breathing to day 28, VFDs will be counted from the end of the last period of assisted breathing to day 28.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants
  0 day | 36 | 27
  1-9 days | 6 | 4
  10-15 days | 3 | 1
  15-19 days | 6 | 12
  20-24 days | 6 | 10
  25-27 days | 2 | 7
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p = 0.02, Regression, Logistic — P-value was given by ordered logistic regression model

7. Secondary Outcome: Duration of Assisted Ventilation Over 28 Days
Description: Duration of assisted ventilation over 28 days in the survivors
Time Frame: 28 days
Population: The analysis was conducted in the subgroup of patients who survived by 6 months.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 35 | 41
days | 22 [9 to 28] | 10 [5 to 20]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Percentage of Patients Achieving Pressure Support Ventilation for 2 Hours
Description: Percentage of patients achieving pressure support ventilation equal to 5 cm H2O with positive end-expiratory pressure (PEEP) equal to 5 cm H2O for 2 hours
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants
  Yes | 25 | 31
  No | 34 | 30
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p = 0.35, Chi-squared

9. Secondary Outcome: Occurrence of Infection
Description: Superficial incisional/wound infections, deep incisional wound infections, and organ/space infections, and ventilator associated pneumonia (all during the 14 days after enrollment)
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants
  Incisional/wound infection | 3 | 1
  Organ/space infection | 1 | 0
  Ventilator associated pneumonia | 20 | 14
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the percentages of patients who developed incision/wound infection events by day 14; Test type: Superiority; p = 0.36, Fisher Exact
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the percentages of patients who developed organ/space infection events by day 14; Test type: Superiority; p = 0.50, Fisher Exact
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the percentages of patients who developed ventilator-associated pneumonia by day 14; Test type: Superiority; p = 0.20, Fisher Exact

10. Secondary Outcome: Occurrence of Thromboembolic Events
Description: Thromboembolic events are measured by ultrasound of the deep venous system or CT-angiography of the chest ordered for clinical purposes/by treating clinicians
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants | 10 | 8
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p = 0.56, Chi-squared — The threshold for statistical significance was p=0.05

11. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Over 7 Days
Description: SOFA score at 3 and 7 days. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems which are added up. Each score ranges from 0 to 4. SOFA score ranges from 0 (best) to 24 (worst).
Time Frame: 7 days
Population: Data were collected in the patients who were still in hospital alive.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
score on a scale
  Day 3: number analyzed (Participants) | 54 | 56
  Day 3 | 9.2 (3.1) | 8.6 (3.1)
  Day 7: number analyzed (Participants) | 47 | 49
  Day 7 | 8.5 (3.8) | 7.7 (4.8)
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the SOFA score between two arms at Day 3; Test type: Superiority; p = 0.32, t-test, 2 sided
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the SOFA score between two arms at Day 7; Test type: Superiority; p = 0.33, t-test, 2 sided

12. Secondary Outcome: Non-pulmonary Sequential Organ Failure Assessment (SOFA) Over 7 Days
Description: Non-pulmonary SOFA score at 3 and 7 days. The score is based on 5 different scores, one each for the cardiovascular, hepatic, coagulation, renal and neurological systems which are added up. Each score ranges from 0 to 4. SOFA score ranges from 0 (best) to 20 (worst).
Time Frame: 7 days
Population: Data were collected in the patients who were still in hospital alive.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
score on a scale
  Day 3: number analyzed (Participants) | 55 | 60
  Day 3 | 6.0 (3.2) | 5.5 (2.9)
  Day 7: number analyzed (Participants) | 52 | 58
  Day 7 | 5.6 (3.5) | 4.8 (3.8)
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for non-pulmonary SOFA scores between the two arms at Day 3; Test type: Superiority; p = 0.39, t-test, 2 sided
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for non-pulmonary SOFA scores between the two arms at Day 7; Test type: Superiority; p = 0.26, t-test, 2 sided

13. Secondary Outcome: All-cause Mortality
Description: All-cause mortality at 14, 28 and 60 days
Time Frame: 60 days
Population: 4 patients were lost of followup up to 60 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants
  14-day mortality | 12 | 8
  28-day mortality: number analyzed (Participants) | 59 | 59
  28-day mortality | 16 | 15
  60-day mortality: number analyzed (Participants) | 58 | 58
  60-day mortality | 21 | 18
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the mortality between two arms at Day 14; Test type: Superiority; p = 0.29, Chi-squared — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the mortality between the two arms at Day 28; Test type: Superiority; p = 0.83, Chi-squared
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis is for the mortality between the two arms at Day 60; Test type: Superiority; p = 0.56, Chi-squared

14. Secondary Outcome: Glasgow Outcome Score (GCS)
Description: Glasgow Outcome Score at hospital discharge. The GCS is a scale to evaluate level of consciousness in patients with acute brain injury. The scale assesses 3 functions: Eye Opening, Verbal Response, and Motor Response. GCS scores range from 15 (best) to 3 (worst)
Time Frame: 60 days
Population: 11 patients did not have recorded Glasgow Coma Scores at hospital discharge, all of them were expired.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 53 | 56
score on a scale | 10.6 (5.6) | 11.5 (5.3)
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p = 0.41, t-test, 2 sided

15. Secondary Outcome: Plasma Angiopoietin-2
Description: Change in levels of plasma angiopoietin-2 from baseline at 6, 24, 48 and 72 hours since the initiation of the study product infusion.
Time Frame: 72 hours
Population: Plasma samples were not collected due to institutional policies during COVID-19 pandemic, or not available at the required timepoints (e.g. discharged from hospital or death).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 hour: number analyzed (Participants) | 38 | 37
  6 hour | 125 [-807 to 1014] | 184 [-99 to 635]
  24 hour: number analyzed (Participants) | 42 | 44
  24 hour | 407 [-1093 to 1733] | 288 [-966 to 1895]
  48 hour: number analyzed (Participants) | 41 | 43
  48 hour | 879 [-200 to 2514] | 343 [-2622 to 2035]
  72 hour: number analyzed (Participants) | 40 | 44
  72 hour | 594 [-1144 to 2318] | 544 [-3359 to 2219]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma angiopoietin-2 changes from the baseline between two arms at 6 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma angiopoietin-2 changes from the baseline between two arms at 24 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma angiopoietin-2 changes from the baseline between two arms at 48 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma angiopoietin-2 changes from the baseline between two arms at 72 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Plasma Receptor for Advanced Glycation Endproducts (RAGE)
Description: Change in levels of plasma RAGE from baseline at 6, 24, 48 and 72 hours since the initiation of the study product infusion.
Time Frame: 72 hours
Population: Samples were not collected due to the intuitional policies regarding the biospecimen collection during COVID-19 pandemic, or not available at the required timepoint of collection (e.g. hospital discharge, death).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 Hour: number analyzed (Participants) | 38 | 37
  6 Hour | 62 [-839 to 954] | -137 [-1412 to 626]
  24 Hour: number analyzed (Participants) | 42 | 44
  24 Hour | -1249 [-4152 to 598] | 100 [-1712 to 2224]
  48 Hour: number analyzed (Participants) | 41 | 43
  48 Hour | -1603 [-4710 to -338] | -906 [-3945 to 806]
  72 Hour: number analyzed (Participants) | 40 | 44
  72 Hour | -2619 [-8478 to -993] | -2054 [-6275 to -198]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma RAGE changes from the baseline between two arms at 6 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma RAGE changes from the baseline between two arms at 24 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma RAGE changes from the baseline between two arms at 48 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma RAGE changes from the baseline between two arms at 72 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Plasma Interleukin-6 (IL-6)
Description: Change in levels of plasma interleukin-6 from baseline compared to 6, 24, 48 and 72 hours
Time Frame: 72 hours
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 Hour: number analyzed (Participants) | 38 | 37
  6 Hour | -10.1 [-53.0 to 6.9] | -3.3 [-16.5 to 4.3]
  24 Hour: number analyzed (Participants) | 42 | 44
  24 Hour | -9.1 [-60.9 to 19.2] | 5.2 [-12.4 to 82.7]
  48 Hour: number analyzed (Participants) | 41 | 43
  48 Hour | -10.7 [-66.2 to 31.6] | 4.1 [-16.3 to 64.5]
  72 Hour: number analyzed (Participants) | 40 | 44
  72 Hour | -11.7 [-90.3 to 56.6] | 2.8 [-56.0 to 35.5]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-6 changes from the baseline between two arms at 6 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-6 changes from the baseline between two arms at 24 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-6 changes from the baseline between two arms at 48 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-6 changes from the baseline between two arms at 72 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Plasma Interleukin-8 (IL-8)
Description: Change in levels of plasma interleukin-8 from baseline at 6, 24, 48 and 72 hours since the initiation of study product infusion.
Time Frame: 72 hours
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 Hour: number analyzed (Participants) | 38 | 37
  6 Hour | -1.0 [-5.5 to 5.4] | -0.4 [-4.2 to 3.4]
  24 Hour: number analyzed (Participants) | 42 | 44
  24 Hour | -0.3 [-9.0 to 6.8] | 0.3 [-4.9 to 7.3]
  48 Hour: number analyzed (Participants) | 41 | 43
  48 Hour | -2.5 [-4.9 to 4.7] | -0.7 [-5.9 to 3.7]
  72 Hour: number analyzed (Participants) | 40 | 44
  72 Hour | 0.4 [-4.1 to 4.9] | 1.4 [-6.9 to 11.2]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-8 changes from the baseline between two arms at 6 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-8 changes from the baseline between two arms at 24 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-8 changes from the baseline between two arms at 48 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Plasma IL-8 changes from the baseline between two arms at 72 hours since the initiation of the study product infusion; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Plasma Tumor Necrosis Factor Receptor 1 (TNFR-1)
Description: Change in levels of plasma TNFR-1 from baseline at 6, 24, 48 and 72 hours since the initiation of study product infusion.
Time Frame: 72 hours
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 Hour: number analyzed (Participants) | 38 | 37
  6 Hour | -1 [-679 to 734] | 271 [-345 to 1629]
  24 Hour: number analyzed (Participants) | 42 | 44
  24 Hour | 231 [-422 to 2009] | 1047 [294 to 2730]
  48 Hour: number analyzed (Participants) | 41 | 43
  48 Hour | 721 [-517 to 1756] | 1596 [354 to 5821]
  72 Hour: number analyzed (Participants) | 40 | 44
  72 Hour | 382 [-40 to 1438] | 985 [-137 to 2999]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of TNFR-1 at 6 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of TNFR-1 at 24 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of TNFR-1 at 48 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of TNFR-1 at 72 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Plasma Protein C
Description: Change in levels of plasma protein C from baseline at 6, 24, 48 and 72 hours since the initiation of study product infusion.
Time Frame: 72 hours
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 Hour: number analyzed (Participants) | 37 | 36
  6 Hour | 7.3 [-26.1 to 38.7] | -2.9 [-17.0 to 15.0]
  24 Hour: number analyzed (Participants) | 41 | 43
  24 Hour | 8.5 [-8.2 to 27.5] | 6.8 [-27.6 to 30.3]
  48 Hour: number analyzed (Participants) | 40 | 42
  48 Hour | 14.0 [-14.2 to 47.2] | 12.7 [-19.7 to 38.2]
  72 Hour: number analyzed (Participants) | 39 | 43
  72 Hour | 26.7 [-15.3 to 55.6] | 8.3 [-25.3 to 49.1]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of Protein C at 6 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of Protein C at 24 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of Protein C at 48 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of Protein C at 72 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Plasma Angiopoietin-1 (ANG-1)
Description: Change in levels of plasma angiopoietin-1 from the baseline to 6, 24, 48 and 72 hours since the initiation of study product infusion.
Time Frame: 72 hours
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
pg/mL
  6 Hour: number analyzed (Participants) | 38 | 37
  6 Hour | -224 [-1548 to 1799] | -292 [-1366 to 1915]
  24 Hour: number analyzed (Participants) | 42 | 44
  24 Hour | 786 [-8 to 3645] | 582 [-1350 to 1827]
  48 Hour: number analyzed (Participants) | 41 | 43
  48 Hour | 612 [-2033 to 3005] | 661 [-881 to 3977]
  72 Hour: number analyzed (Participants) | 40 | 44
  72 Hour | 148 [-2462 to 3950] | 59 [-1646 to 2557]
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of ANG-1 at 6 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of ANG-1 at 24 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of ANG-1 at 48 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; The analysis for the changes of ANG-1 at 72 hours since the initiation of study product infusion from the baseline; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Plasma Lipoxin A4
Description: Change in levels of plasma lipoxin A4 from baseline compared to 6, 24, 48 and 72 hours
Time Frame: 72 hours
Population: The majority of plasma samples were collected but some were not due to institutional policies on biospecimen collection during COVID-19 pandemic or because patients were no longer available (e.g. discharge, death). Plasma lipoxin A4 levels were not tested because the method depends on a complicated assay that is not validated for human use and is therefore unreliable. As a result, these samples have not been analyzed and will not be analyzed in the future.
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Plasma Resolvin D1
Description: Change in levels of plasma Resolvin D1 from baseline compared to 6, 24, 48 and 72 hours
Time Frame: 72 hours
Population: The majority of plasma samples were collected but some were not due to institutional policies on biospecimen collection during COVID-19 pandemic or because patients were no longer available (e.g. discharge, death). Plasma resolvin D1 levels were not tested because the method depends on a complicated assay that is not validated for human use and is therefore unreliable. As a result, these samples have not been analyzed and will not be analyzed in the future.
Arm/Group | Cell Reconstitution Media | Human Mesenchymal Stromal Cells
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Plasma Keratinocyte Growth Factor (KGF)
Description: Change in levels of plasma KGF from baseline at 6, 24, 48 and 72 hours since the initiation of study product infusion.
Time Frame: 72 hours
Population: Most plasma samples were collected but some were not due to institutional restriction during the COVID-19 pandemic or patient unavailable (e.g. discharge, death). KGF doesn't accurately reflect biological activity of the mesenchymal stromal cell (MSC) treatment, and KGF assay is unreliable for determining the quantity released by MSCs (the therapeutic product) versus the release from endogenous cells within the patient. Thus, KGF levels have not been analyzed and will not analyzed in the future.
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Urine Microalbumin
Description: Change in levels of urine microalbumin from baseline compared to 24 and 48 hours
Time Frame: 48 hours
Population: The majority of urine samples were collected, but some were not due to institutional policies on biospecimen collection during the COVID-19 pandemic or because patients were no longer available (e.g., discharge, death). However, this measurement isn't reliable, as it doesn't accurately reflect kidney function or correlate intelligently with the effects of MSC therapy on kidney function. As a result, urine microalbumin levels were not analyzed and will not analyzed in the future.
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Total Protein in Min-bronchoalveolar Lavage (mBAL)
Description: Change in total protein levels in from baseline to day 2
Time Frame: 2 days
Population: The mini-BAL samples were not able to be collected during the COVID-19 pandemic due to local COVID policies and safety concerns. Collecting bronchoalveolar (BAL) samples would have been a major risk for spreading the COVID-19 virus to health care workers.
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Tolerability of the hMSCs - Incidence of Pre-specified Infusion-associated Events and Unexpected Severe Adverse Events
Description: Tolerability of the hMSCs, defined as the incidence of pre-specified infusion-associated events and unexpected severe adverse events in ARDS patients treated with human MSCs
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
Number analyzed (Participants) | 59 | 61
Participants | 2 | 2
Statistical Analysis 1: Comparison: Human Mesenchymal Stromal Cells vs Cell Reconstitution Media; Test type: Superiority; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through 28 days from study product infusion. Death data was collected up to 6 months.
Arm/Group | Human Mesenchymal Stromal Cells | Cell Reconstitution Media
All-Cause Mortality (participants affected / at risk) | 24/59 | 21/61
Serious Adverse Events (participants affected / at risk) | 3/59 | 2/61
Other Adverse Events (participants affected / at risk) | 9/59 | 6/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Mesenchymal Stromal Cells (N=59) | Cell Reconstitution Media (N=61)
ECMO (Cardiac disorders) | 1 (1) | 0 (0)
Asymmetric perfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Partial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Tension pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PEA arrest (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Mesenchymal Stromal Cells (N=59) | Cell Reconstitution Media (N=61)
Deep Vein Thrombosis (Nervous system disorders) | 3 (3) | 2 (2)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
VAP Sepsis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decrease in oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
C, diff infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diplopia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03818854/Prot_001.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03818854/SAP_002.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03818854/ICF_000.pdf